CLINICAL TRIAL: NCT02735668
Title: Is Multimodal Physiotherapy More Effective Than Exercise Alone in Women With Peripheral Persistent Pain Following Breast Cancer Treatment? A Single-blinded Randomized Clinical Trial
Brief Title: Physiotherapy in Women With Peripheral Persistent Pain Following Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Virginia Prieto Gómez, Research Expert of Healthcare (Msc), University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPSM_UAH_VPG
Record Dates: First submitted 2016-04-03; First posted 2016-04-13 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Pain; Breast Cancer
Keywords: Shoulder Pain; Pattern Motor; Physical Therapy Modalities; Breast Cancer Treatment
MeSH Terms: conditions — Shoulder Pain; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Shoulder Conventional Exercises (Active Comparator): The protocol consists in:
  * Flexibility and Strengthening Exercises of the shoulder muscles conventionally performed in shoulder pathology treatment.
  * Therapeutic Education about chronic shoulder pain.
  The treatment duration is 1 day per week during 6 weeks.
  Interventions: Other: Shoulder Conventional Exercises; Behavioral: Therapeutic Education
- Multimodal Physiotherapy (Experimental): The protocol consists in:
  * Dry Needling in active myofascial trigger points.
  * Neurodynamic techniques.
  * Scapular exercises.
  * Therapeutic Education about chronic shoulder pain.
  The treatment duration is 1 day per week during 6 weeks.
  Interventions: Other: Multimodal Physiotherapy; Other: Scapular exercises; Behavioral: Therapeutic Education
- Scapular exercises (Experimental): The protocol consists in:
  * Scapular exercises
  * Therapeutic Education about chronic shoulder pain.
  The treatment duration is 1 day per week during 6 weeks.
  Interventions: Other: Scapular exercises; Behavioral: Therapeutic Education

INTERVENTIONS:
Other: Shoulder Conventional Exercises — The protocol consists in:
  • Flexibility and Strengthening Exercises of the shoulder muscles conventionally performed in shoulder pathology treatment:
  * Mobilisation Joint Exercises.
  * Isometrics and Resisted Exercises (elastic bands).
  Other Names: Conventional physical therapy
  Arms: Shoulder Conventional Exercises
Other: Multimodal Physiotherapy — The protocol consists in:
  * Dry Needling in active myofascial trigger points related to shoulder joint (optimal hygiene and disinfection before and after needling). Special care in muscles located in the arm in women with axillary node dissection.
  * If Upper Limb Neural Tension Test is positive, neurodynamic techniques will be included.
  Other Names: Specific physical therapy
  Arms: Multimodal Physiotherapy
Other: Scapular exercises — The protocol consists in:
  Scapula-focused exercises: based on evaluation of scapular dyskinesis and Kinetic Medial Rotation Test as well as inherent characteristics of each woman, individualized scapular exercises were prescribed based on a motor control approach with emphasis on obtaining a neutral scapular orientation.
  Other Names: Specific physical therapy
  Arms: Multimodal Physiotherapy; Scapular exercises
Behavioral: Therapeutic Education — The protocol consists in:
  Therapeutic Education about chronic shoulder pain using a slide show, anatomical models, providing information and analysis of real clinical cases.
  Other Names: Hygienic and behavioral advises

SUMMARY:
The aim of this study is to determine the effectiveness of a multimodal physiotherapy intervention including scapula exercises in addition to deep dry needling and neurodynamic techniques versus scapula exercises only versus conventional shoulder exercises on pain intensity, perceived disability, scapula muscle activity and health-related quality of life.

DETAILED DESCRIPTION:
Introduction: chronic shoulder pain is a frequent consequence after breast cancer treatment with a reported prevalence of 25% to 60% and is commonly termed "Persistent Pain after Breast Cancer Treatment" (PPBCT). Frequently, PPBCT includes neuropathic pain due to damage of neural tissue during surgery. However, recent studies, consider that myofascial pain syndrome and heightened mechanosensitivity of neural tissue can be also present in this women. Although PPBCT is typically managed with pharmacological treatment,currently, physiotherapy is presented as an alternative method. Physiotherapy in relation to the shoulder, commonly, focuses its treatment with therapeutic exercise. In this sense, there is great controversy about which are the most appropriate exercises. Recent authors, bet for more precise and analytical exercises in relation with scapula and reject conventional exercises for the shoulder. Taking into account each of the sources of pain presented by these women and the benefits of therapeutic exercise, it would be interesting to study which approach of physiotherapy treatment would be more appropriate in these women.

Subjects and methods: A randomized clinical trial, the examiner being blinded unaware of the intervention group to which subjects were assigned. Participants will be randomly assigned to three groups:

An experimental group, where the participants will be treated with Multimodal Physiotherapy;

Another experimental group where will be realized Scapular Exercises only;

And a third group where will be done Shoulder Conventional Exercises.

Pre- intervention, immediate post-intervention, 3, and 6 months assessments will be made. The selection criteria will be: women with peripheral persistent pain following breast cancer treatment (surgery and/or radiotherapy and/or chemotherapy) with pain for at least 6 months. The participants must understand and sign freely Informed Consent.

Sample size: 30 women for each group.

Data Analysis: A descriptive analysis of all variables will be performed. It will be established for all cases a confidence level of 95% (p <0.05). The effectiveness will be assessed by comparing the experienced change of the three goups in outcome variables between physicaltherapy examinations.

ELIGIBILITY:
Inclusion Criteria:

* Women with peripheral persistent pain following breast cancer treatment (surgery and/or radiotherapy and/or chemotherapy) with pain for at least 6 months.
* Women who do not present contraindications for physiotherapy (infection, metastasis, locoregional recurrence).
* Women who have read, understood and signed informed consent freely

Exclusion Criteria:

* Women treated with bilateral breast cancer.
* Women with shoulder pain episodes prior to breast cancer treatment.
* Women with predominant central sensitization pain identified by the Central Sensitization Inventory (> 40 points)
* Women with cognitive limitations to understand the information provided, instructions for treatment and consent to their participation in the study.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change from baseline VAS at after 9 physical therapy sessions, 3 and 6 months after baseline assessments will be require
  Visual analogue scale (VAS).100 mm horizontal with pain descriptors marked "no pain" on the left side or "worst imaginable pain".

SECONDARY OUTCOMES:
Pain and Disability | At baseline, after 9 physical therapy sessions, 3 and 6 months after baseline assessments were required.
  The questionnaire Shoulder Pain and Disability Index validated in Spanish, to measure the intensity and information on the characteristics of pain and the level of shoulder disability is used. This questionnaire contains a numerical scale from 0 to 10 to collect each answer.
Root-Mean-Square (RMS) EMG Amplitude | At baseline, after 9 physical therapy sessions, 3 and 6 months after baseline assessments were required.
  Quantification of motor unit recruitment (electrical activity), by analyzing the RMS, expressed in microvolts (normalized data expressed as a percentage) of the muscles: upper and lower trapezius, middle deltoid, infraspinatus and serratus anterior during Abduction Movement
Onset EMG | At baseline, after 9 physical therapy sessions, 3 and 6 months after baseline assessments were required.
  Beginning of motor activation, expressed in seconds (s), of the muscles: upper and lower trapezius, middle deltoid, infraspinatus and serratus anterior during Abduction Movement.
Health-related quality of life | At baseline, after 9 physical therapy sessions, 3 and 6 months after baseline assessments were required.
  Questionnaire: Assessment of Cancer Therapy-Breast (FACT-B) Spanish version 4
Myofascial Pain Syndrome. Active myofascial trigger points of the muscles involved in shoulder. Travell and Simon's Criteria were used. | At baseline, after 9 physical therapy sessions, 3 and 6 months after baseline assessments were required.
  Travell and Simon's Criteria consists in (Wolfe et al 1992):
  The major criteria include:
  1. A patient's regional pain complaint;
  2. Palpation of a trigger point elicits a stereotypic zone of referred pain specific to that muscle;
  3. Identification of a palpable taut band;
  4. As well as a palpable, and exquisitely tender spot along the length of that taut band;
  5. Some degree of restricted range of motion of the involved muscle.
  Three minor criteria have been suggested to further aid in the diagnosis of myofascial pain syndrome:
  1. Palpation of a trigger point should reproduce the clinical pain complaint;
  2. A local twitch response may be elicited by transverse snapping or needling of the trigger point;
  3. The alleviation of pain by trigger point inactivation.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia P Gómez, PhD Student, Principal Investigator — Department of Physiotherapy. University of Alcala.
Locations (1):
- Teacher care and research in physiotherapy Unit. Department of Physiotherapy. University of Alcala., Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No